CLINICAL TRIAL: NCT01867047
Title: Effects of Angiotensin Converting Enzyme Inhibitors on Total Hip and Knee Arthroplasty Patients
Brief Title: ACE-Inhibitor Effects on Total Hip and Knee Arthroplasty Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Following an interim analysis the study team felt that there was enough data that showed no significant difference.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00037620; Pro00037620 (Other: Duke University IRB)
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Results first posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-06

CONDITIONS: Adverse Effects of Angiotensin-converting-enzyme Inhibitors; Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuation Group (Experimental): Subjects randomized to this group will continue their ACE-I through the day of surgery
  Interventions: Drug: ACE-I Continuation group
- Cessation Group (Experimental): Subjects randomized to this group will stop their ACE-I two days prior to surgery (last dose >48 hours prior to surgery)
  Interventions: Drug: ACE-I Cessation group

INTERVENTIONS:
Drug: ACE-I Cessation group — Subjects stop ACE-I 48 hours prior to surgery. Examples of possible ACE-I drugs include:
  benazepril (Lotensin), captopril (Capoten), enalapril (Vasotec, Epaned), fosinopril (Monopril), lisinopril (Prinivil, Zestril), moexipril (Univasc), perindopril (Aceon), quinapril (Accupril), ramipril (Altace), trandolapril (Mavik)
  Arms: Cessation Group
Drug: ACE-I Continuation group — Subjects take ACE-I through day of surgery. Examples of possible ACE-I drugs include:
  benazepril (Lotensin), captopril (Capoten), enalapril (Vasotec, Epaned), fosinopril (Monopril), lisinopril (Prinivil, Zestril), moexipril (Univasc), perindopril (Aceon), quinapril (Accupril), ramipril (Altace), trandolapril (Mavik)
  Arms: Continuation Group

SUMMARY:
The purpose of this study is to determine the effects of Angiotension Converting Enzyme Inhibitors (ACE-I) during surgery and in the immediate postoperative period for patients undergoing elective total hip or knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients electing to undergo primary or revision total hip or knee arthroplasty
* Currently taking an ACE-I

Exclusion Criteria:

* Trauma patients
* Immunosuppressed patients (HIV/AIDS, organ transplant recipients, chemotherapy patients, chronic steroid use)
* Patients with history of severe hypertension related illness such as hypertension associated with stroke or myocardial infarction
* Patients in who continuation of their ACE-I is expressly mandated by their prescribing physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06-24 (Actual); Study Completion 2016-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bolognesi, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were prescreened by the study team and then identified and presented to the surgeon during the preoperative clinic visit. Once IRB approval was granted on 8-9-2012 study team started screening the clinic schedule for potential participants.
Pre-assignment Details: Randomization of participants occurred only if the proposed inclusion/exclusion criteria were met.
Groups:
- Continuation Group: ACE-I Continuation group: Subjects take ACE-I through day of surgery
- Cessation Group: ACE-I Cessation group: Subjects stop ACE-I 48 hours prior to surgery
Period: Overall Study
Arm/Group | Continuation Group | Cessation Group
Started | 31 | 28
Completed | 23 | 23
Not Completed | 8 | 5
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 2 | 0
Not completed — surgery not indicated in protocol | 1 | 2

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuation Group | Cessation Group | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 13 | 29
  >=65 years | 7 | 10 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (10.8) | 63.7 (8.7) | 63.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 15 | 12 | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Mild Hypotension
Description: The number of participants with mild hypotension (Systolic Blood Pressure (SBP) less than 85 mmHG) will be recorded.
Time Frame: From baseline to discharge from hospital (approximately 5 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation Group | Cessation Group
Number analyzed (Participants) | 23 | 23
Participants
  Intraoperative | 14 | 9
  Postoperative | 3 | 2
Statistical Analysis 1: Comparison: Continuation Group vs Cessation Group; Statistical analysis for intraoperative mild hypotension; Test type: Superiority; p = 0.140, t-test, 2 sided
Statistical Analysis 2: Comparison: Continuation Group vs Cessation Group; Statistical analysis for postoperative mild hypotension; Test type: Superiority; p = 1.000, t-test, 2 sided

2. Primary Outcome: Number of Participants With Severe Hypotension
Description: The number of participants with severe hypotension (Systolic Blood Pressure less than 65 mmHG) will be recorded.
Time Frame: From baseline to discharge from hospital (approximately 5 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation Group | Cessation Group
Number analyzed (Participants) | 23 | 23
Participants
  Intraoperative | 1 | 0
  Postoperative | 0 | 0

3. Primary Outcome: Number of Participants Given Vasopressors
Description: The number of participants who received vasopressors.
Time Frame: Discharge from hospital (approximately 5 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation Group | Cessation Group
Number analyzed (Participants) | 23 | 23
Participants
  Intraoperative | 19 | 14
  Postoperative | 0 | 0
Statistical Analysis 1: Comparison: Continuation Group vs Cessation Group; Analysis for number of participants given vasopressors intraoperatively; Test type: Superiority; p = 0.102, t-test, 2 sided

4. Secondary Outcome: Number of Participants Transferred to Intensive Care Unit (ICU)
Description: The number of participants transferred to Intensive Care Unit (ICU) will be recorded
Time Frame: Discharge from hospital (approximately 5 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation Group | Cessation Group
Number analyzed (Participants) | 23 | 23
Participants | 1 | 0

5. Secondary Outcome: Number of Participants That Received Allogeneic Blood
Description: The number of participants that received allogeneic blood will be recorded.
Time Frame: Discharge from hospital (approximately 5 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation Group | Cessation Group
Number analyzed (Participants) | 23 | 23
Participants | 1 | 0

6. Secondary Outcome: Number of Participants With Acute Kidney Injury
Description: Number of participants with acute kidney injury will be recorded.
Time Frame: Discharge from hospital (approximately 5 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation Group | Cessation Group
Number analyzed (Participants) | 23 | 23
Participants | 5 | 3
Statistical Analysis 1: Comparison: Continuation Group vs Cessation Group; Test type: Superiority; p = 0.700, t-test, 2 sided

7. Post Hoc Outcome: Length of Stay
Description: Length of stay in days
Time Frame: Discharge from hospital (approximately 5 days)
Measure: Median (Full Range); unit: Days
Groups:
- Continuation Group: Subjects randomized to this group will continue their ACE-I through the day of surgery
  ACE-I Continuation group: Subjects take ACE-I through day of surgery. Examples of possible ACE-I drugs include:
  benazepril (Lotensin), captopril (Capoten), enalapril (Vasotec, Epaned), fosinopril (Monopril), lisinopril (Prinivil, Zestril), moexipril (Univasc), perindopril (Aceon), quinapril (Accupril), ramipril (Altace), trandolapril (Mavik)
- Cessation Group: Subjects randomized to this group will stop their ACE-I two days prior to surgery (last dose >48 hours prior to surgery)
  ACE-I Cessation group: Subjects stop ACE-I 48 hours prior to surgery. Examples of possible ACE-I drugs include:
  benazepril (Lotensin), captopril (Capoten), enalapril (Vasotec, Epaned), fosinopril (Monopril), lisinopril (Prinivil, Zestril), moexipril (Univasc), perindopril (Aceon), quinapril (Accupril), ramipril (Altace), trandolapril (Mavik)
Arm/Group | Continuation Group | Cessation Group
Number analyzed (Participants) | 23 | 23
Days | 2.0 [1 to 13] | 2.0 [1 to 7]
Statistical Analysis 1: Comparison: Continuation Group vs Cessation Group; Test type: Superiority; p = 0.702, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Baseline to hospital discharge (approximately 5 days)
Description: The study team only collected adverse events that were unanticipated and reported to the study coordinator.
Arm/Group | Continuation Group | Cessation Group
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

LIMITATIONS AND CAVEATS:
Limitations of this study include a low power, as the investigators assessed a relatively small number of participants, and as such the investigators recommend repeated studies with larger numbers of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes